CLINICAL TRIAL: NCT05481437
Title: Specified Drug Use Surveillance for ADCETRIS Intravenous Infusion 50 mg -Untreated CD30 Positive Hodgkin Lymphoma (Pediatric)
Brief Title: A Survey of Brentuximab Vedotin in Pediatric Participants With Hodgkin Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brentuximab-5019; jRCT2031220244 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brentuximab Vedotin: Participants will receive Brentuximab Vedotin injection 50 mg once every 2 weeks and AVD treatment (doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine).
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin injection, 50 mg, once every 2 weeks
  Other Names: ADCETRIS Intravenous Infusion

SUMMARY:
This study is a survey in Japan of Brentuximab Vedotin used to treat children or teenagers with Hodgkin lymphoma (HL). The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from Brentuximab Vedotin especially myelosupression, peripheral neuropathy, and lung disorder.

During the study, pediatric participants with HL will take Brentuximab Vedotin injection and AVD treatment (doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine) according to their clinic's standard practice. The study doctors will check for side effects from Brentuximab Vedotin for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naive participants
2. CD30 positive participants
3. Participants treated with the study drug in combination with doxorubicin hydrochloride, vinblastine sulfate, and dacarbazine (AVD).
4. Participants aged < 18 years at the start of this drug.

Exclusion Criteria:

Participants with contraindications to the study drug.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Experienced Myelosuppression | Up to 26 Weeks
Percentage of Participants who Experienced Peripheral Neuropathy | Up to 26 Weeks
Percentage of Participants who Experienced Lung Disorder | Up to 26 Weeks

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Event (AE) Leading to Brentuximab Vedotin Discontinuation, Serious Adverse Event (SAE), and Grade 3 or Higher Adverse Event (AE) | Up to 26 Weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product. An adverse event does not necessarily have a causal relationship with the intervention. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity grades will be evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE). Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately lifethreatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Percentage of Participants Who Achieve or Maintain Any Best Response | Up to 26 Weeks
  Best response is defined as the cumulative numbers of participants who achieve each level of best response including complete response (CR), complete response/unconfirmed (CRu), partial response (PR), Stable Disease (SD), Progressive Disease (PD) and Relapsed Disease (RD) after treatment. Best response will be assessed by International Working Group (IWG) criteria or Antitumor effect assessment criteria for pediatric HL of Japan Childhood Leukemia and Lymphoma Study Group (JPLSG) version.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/9bb9378e41504b5a